CLINICAL TRIAL: NCT07316179
Title: A Prospective Observational Study Comparing the El Ganzouri Risk Index and Airway Ultrasonography in Predicting Difficult Intubation in Patients Undergoing Bariatric Surgery
Brief Title: Predicting Difficult Intubation in Bariatric Surgery: Comparison of El Ganzouri Risk Index and Airway Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10/9
Record Dates: First submitted 2025-11-20; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Obesity & Overweight; Obesity Difficult Airway Airway Management; Obesity (Disorder); Difficult Airway; Difficult Intubation in Obesity; Difficult Laryngoscopy
Keywords: El Ganzouri Risk Index; Difficult airway; Obesity; Airway Ultrasonography; Airway Management
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed as a prospective observational study and will be conducted at the Health Sciences University Antalya Training and Research Hospital. Adult patients scheduled to undergo bariatric surgery will be included.

The aim of this study is to compare the El Ganzouri Risk Index (EGRI) and airway ultrasonography (USG) parameters in predicting difficult intubation and to evaluate their relationship with the Cormack-Lehane (CL) score obtained during direct laryngoscopy.

Before surgery, each participant will be evaluated using both the EGRI scoring system and airway USG. During general anesthesia, tracheal intubation will be performed using direct laryngoscopy, and data including the CL score, intubation time, number of attempts, and the need for videolaryngoscopy will be recorded based on the anesthesiologist's observations.

The collected data will be analyzed by classifying participants according to the presence or absence of difficult intubation, and statistical comparisons will be performed between EGRI scores and airway ultrasonography parameters. The results of this study may contribute to improved preoperative airway assessment and enhanced patient safety in bariatric surgery.

DETAILED DESCRIPTION:
Background and Rationale

Airway management is a fundamental aspect of anesthesia practice and plays a critical role in ensuring patient safety during surgical procedures. Under general anesthesia, suppression of spontaneous breathing necessitates the secure maintenance of airway patency. Successful tracheal intubation is essential for the safe conduct of surgery; however, in some patients, intubation may be unexpectedly difficult. According to current definitions, difficult intubation is characterized by the inability to adequately visualize glottic structures using standard techniques, resulting in failure or the need for multiple attempts. Delayed or failed intubation following anesthesia induction can lead to serious complications, including hypoxemia, aspiration, bradycardia, and cardiac arrest. Therefore, accurate preoperative prediction of difficult intubation is of critical importance. Early identification of difficult airway cases allows for timely implementation of alternative techniques and airway devices, thereby reducing perioperative risks and complications.

Obesity has emerged as a major global health concern and represents a significant risk factor for difficult intubation. Bariatric surgery is indicated in individuals with a body mass index (BMI) ≥40 kg/m² or ≥35 kg/m² in the presence of serious comorbidities, with the aim of reducing obesity-related metabolic, cardiovascular, and respiratory complications while improving quality of life. However, obese patients present unique challenges in airway management due to increased adipose tissue in the neck, reduced cervical-pharyngeal angles, and enlarged soft tissue structures. These anatomical factors impair visualization of laryngeal structures and may prolong intubation time, thereby increasing the risk of airway-related complications.

EGRI was developed as a comprehensive scoring system for predicting difficult intubation by incorporating multiple airway assessment parameters, including mouth opening, Mallampati classification, neck mobility, mandibular protrusion, upper incisors, thyromental distance, and a history of difficult intubation. Several studies have demonstrated the clinical utility and predictive value of EGRI in preoperative airway assessment.

Airway USG has recently gained attention as a non-invasive method for predicting difficult intubation. This technique enables real-time visualization of airway anatomy and allows measurement of parameters such as skin-to-epiglottis distance, skin-to-hyoid bone distance, skin-to-vocal cord distance, and tongue thickness. Previous studies suggest that USG may provide predictive accuracy comparable to or greater than that of traditional clinical indices, including EGRI. However, evidence regarding its use in patients undergoing bariatric surgery remains limited, underscoring the need for further investigation.

Direct laryngoscopy remains the standard technique for airway visualization during tracheal intubation. CL grading system, which ranges from Grade I (full view of the glottis) to Grade IV (no visible glottic structures), provides an objective assessment of intubation difficulty. In this study, CL score will be used as a reference standard to compare the predictive performance of EGRI and airway USG parameters in participants undergoing bariatric surgery.

Study Objectives

Patients scheduled for bariatric surgery are at increased risk of difficult intubation, necessitating the use of accurate and objective preoperative assessment tools. Traditional clinical scoring systems, such as EGRI, are practical and widely used; however, their predictive accuracy may be limited by subjectivity. Airway USG is an emerging, non-invasive technique that provides direct visualization of airway structures, but further investigation is required to establish its role in this patient population.

The primary objective of this study is to compare the predictive performance of EGRI and airway USG parameters in identifying difficult intubation in participants with obesity undergoing bariatric surgery. A secondary objective is to evaluate the association between preoperative airway assessment findings and intraoperative CL scores obtained during direct laryngoscopy.

By determining which assessment method demonstrates greater accuracy and reliability, this study aims to generate evidence that may contribute to improved preoperative airway evaluation and enhanced patient safety in bariatric surgery.

Study Design

This study is designed as a prospective observational clinical study. The primary aim is to compare EGRI and airway USG parameters in predicting difficult intubation in adult participants scheduled for bariatric surgery and to evaluate their association with CL scores obtained during direct laryngoscopy.

During the preoperative period, all participants will undergo airway assessment using both the EGRI scoring system and airway USG. Tracheal intubation will be performed under general anesthesia using direct laryngoscopy. The degree of intubation difficulty will be documented based on the anesthesiologist's observations, including CL grade, intubation time, and number of intubation attempts.

The collected data will be classified according to the presence or absence of difficult intubation. Statistical analyses will be performed to compare the predictive performance of EGRI scores and airway USG parameters and to evaluate their relationship with direct laryngoscopic findings.

Data Analysis

Data will be analyzed using appropriate statistical software. Participants will be categorized into two groups based on the presence or absence of difficult intubation, as determined by intraoperative findings.

Descriptive statistics will be used to summarize demographic and clinical characteristics. Continuous variables will be reported as mean ± standard deviation or median with interquartile range, depending on data distribution. Categorical variables will be presented as frequencies and percentages.

Appropriate statistical tests will be applied to compare EGRI scores and airway USG parameters between groups. Correlation analyses will be performed to evaluate the relationships among preoperative airway USG measurements, EGRI scores, and intraoperative CL grades.

The diagnostic performance of EGRI scores and airway USG parameters in predicting difficult intubation will be assessed using comparative statistical methods.

A p-value of <0.05 will be considered statistically significant.

Expected Outcomes

Primary Outcome:

To compare the diagnostic effectiveness of EGRI and airway USG parameters in predicting difficult intubation in adult participants scheduled to undergo bariatric surgery.

Secondary Outcome

To evaluate the association between EGRI scores and airway USG measurements and clinical variables, including intubation time, number of intubation attempts, and the occurrence of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 to 65 years.
* ASA physical status classification II or III.
* Scheduled to undergo elective bariatric surgery under general anesthesia.
* Patients who voluntarily agree to participate in the study and sign the informed consent form.

Exclusion Criteria:

* Patients younger than 18 years or older than 65 years
* Presence of upper airway anatomical pathology
* History of tracheal or thyroid surgery.
* History of radiotherapy to the head and neck region.
* Cervical spine anomalies.

Individuals unwilling to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult participants aged 18 to 65 years with ASA physical status II or III who are scheduled to undergo elective bariatric surgery under general anesthesia. Eligible participants must provide written informed consent prior to inclusion in the study. Participants with upper airway anatomical pathology, previous tracheal or thyroid surgery, head or neck masses, history of radiotherapy to the head and neck region, cervical spine anomalies, or those unwilling to participate will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07-28 (Estimated)

PRIMARY OUTCOMES:
Association between each individual ultrasound parameter and difficult laryngoscopy | Baseline (preoperative period)
  Difficult laryngoscopy will be defined as CL grades III-IV, which will serve as the reference standard. Each predefined airway ultrasonography parameter will be analyzed independently to evaluate its association with difficult laryngoscopy. No composite score will be calculated.
  The following preoperative airway ultrasonography measurements will be assessed individually:
  Tongue base thickness Hyomental distance in the neutral position Hyomental distance in the extended position Hyomental ratio (extension/neutral) Skin-to-hyoid distance Skin-to-epiglottis distance Skin-to-vocal cords (anterior commissure) distance Skin-to-cricoid cartilage distance Pre-epiglottic space depth
  Unit of Measure Centimeters (cm) for all linear measurements

SECONDARY OUTCOMES:
Comparison of Diagnostic Performance Between the EGRI and Airway USG Measurements | Baseline (preoperative period)
  The diagnostic performance of the El Ganzouri Risk Index (EGRI) and individual airway ultrasonography measurements will be compared for the prediction of difficult laryngoscopy.
  The EGRI is a seven-item multivariable bedside airway assessment index with a total score ranging from 0 to 12, where higher scores indicate an increased risk of difficult intubation. Each item is scored using predefined cut-off values and summed to generate a single composite EGRI score.
  The EGRI components include:
  Mouth opening Thyromental distance Mallampati classification Neck extension Mandibular protrusion Body weight History of difficult intubation
  Airway USG parameters will be analyzed independently, as defined in the primary outcome measure. Difficult laryngoscopy will be defined as CL grades III-IV, which will serve as the reference standard.
  Unit of Measure Score (0-12) for the El Ganzouri Risk Index Centimeters (cm) for airway ultrasonography measurements
Association Between Airway Ultrasonography Parameters and Intubation Performance | Perioperative period (during tracheal intubation)
  Associations between individual preoperative airway ultrasonography measurements and intubation performance metrics will be evaluated. Each airway ultrasonography parameter will be analyzed independently.
  Intubation performance metrics include:
  Intubation time Number of intubation attempts Requirement for videolaryngoscopy Occurrence of intubation-related complications
  Unit of Measure Seconds for intubation time Count for number of intubation attempts Binary (yes/no) for videolaryngoscopy requirement Binary (yes/no) for intubation-related complications
Predictive Performance of the EGRI for Difficult Laryngoscopy | Baseline (preoperative period)
  The predictive performance of EGRI total score will be evaluated for the identification of difficult laryngoscopy. Difficult laryngoscopy will be defined as CL grades III-IV, which will serve as the reference standard. The EGRI is a composite bedside airway assessment index with a total score ranging from 0 to 12, where higher scores indicate an increased risk of difficult intubation.
Association Between Early Intraoperative Hemodynamic Instability and Difficult Laryngoscopy | Perioperative period (first 30 minutes of surgery)
  The association between early intraoperative hemodynamic instability and difficult laryngoscopy will be evaluated. Difficult laryngoscopy will be defined as CL grades III-IV, which will serve as the reference standard.
  Hemodynamic parameters will be recorded at 5-minute intervals during the first 30 minutes of surgery, including heart rate, arterial blood pressure, and peripheral oxygen saturation. The following pre-specified derived variables will be used for analysis:
  Lowest mean arterial pressure (MAP) within the first 30 minutes Lowest peripheral oxygen saturation (SpO₂) within the first 30 minutes Duration of hypotension, defined as the number of 5-minute intervals with MAP < 65 mmHg Duration of hypoxemia, defined as the number of 5-minute intervals with SpO₂ < 90% Maximum decrease in MAP from the pre-induction baseline (ΔMAP) Each derived variable will be analyzed as an indicator of hemodynamic instability.
Incidence and Clinical Correlates of Difficult Laryngoscopy in Obese Adults Undergoing Bariatric Surgery | Perioperative period (during tracheal intubation)
  The incidence of difficult laryngoscopy will be determined in adult participants with obesity undergoing bariatric surgery. Difficult laryngoscopy will be defined as CL grades III-IV, which will serve as the reference standard.
  Associations between difficult laryngoscopy and selected demographic and clinical variables, including body mass index (BMI) and sex, will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Tercan, Study Director — University of Health Sciences Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Antalya, Turkey (Türkiye)